CLINICAL TRIAL: NCT01501487
Title: MINT I Multi- Institutional Neo-adjuvant Therapy MammaPrint Project I
Acronym: MINT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Agendia (Industry)
Collaborators: University of South Florida (Other); University of Miami (Other); Morton Plant Mease Health Care (Other); AdventHealth (Other); Plano Cancer Center (Unknown); Ohio State University Comprehensive Cancer Center (Other); University of Oklahoma (Other); University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P0334
Record Dates: First submitted 2011-12-22; First posted 2011-12-29 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; neo adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HER2 negative patients (Active Comparator): In order to provide some consistency in management and have a treatment policy in place only recommended therapy with several well accepted and presumed equivalent chemotherapy regimens will be used. The proposed neo-adjuvant chemotherapy regimens for HER2 negative patients include:
  1. TAC chemotherapy
  2. TC chemotherapy
  3. Dose Dense AC or FEC100 followed by paclitaxel or docetaxel chemotherapy
  Interventions: Drug: TAC chemotherapy; Drug: TC chemotherapy; Drug: Dose Dense AC or FEC100 followed by paclitaxel or docetaxel chemotherapy
- Her2 positive patients (Active Comparator): The proposed neo-adjuvant chemotherapy regimens for HER2 negative patients is TCH chemotherapy.
  Interventions: Drug: TCH chemotherapy; Drug: T + trastuzumab followed by CEF + trastuzumab; Drug: Dose dense AC followed by T + trastuzumab; Drug: Dose dense AC followed by T + trastuzumab + pertuzumab; Drug: PTH followed by dose dense AC of FEC

INTERVENTIONS:
Drug: TAC chemotherapy — Docetaxel 75 mg/m2 IV day 1, Doxorubicin 50 mg/m2 IV day 1, Cyclophosphamide 500 mg/m2 IV day 1; Cycled every 21 days for 6 cycles
  Arms: HER2 negative patients
Drug: TC chemotherapy — Docetaxel 75 mg/m2 IV day 1, Cyclophosphamide 600 mg/m2 IV day 1; Cycled every 21 days for 6 cycles
  Arms: HER2 negative patients
Drug: Dose Dense AC or FEC100 followed by paclitaxel or docetaxel chemotherapy — Doxorubicin 60 mg/m2 IV day 1, Cyclophosphamide 600 mg/m2 IV day 1, Cycled every 14 days for 4 cycles, OR 5-Fluorouracil 500 mg/m2 IV day 1, Epirubicin 100 mg/m2 IV day 1, Cyclophosphamide 500 mg/m2 IV day 1; Cycled every 21 days for 3 cycles Followed by Paclitaxel 80 mg/m2 by 1 h IV infusion weekly for 12 weeks, OR Docetaxel 100mg/m2 IV day 1 cycled every 21 days for 3 or 4 cycles
  Arms: HER2 negative patients
Drug: TCH chemotherapy — Docetaxel 75 mg/m2 IV day 1, followed by Carboplatin AUC 6 IV day 1; Cycled every 21 days for 6 cycles Trastuzumab initial dose of 4 mg/kg over 90 minute IV infusion, then 2 mg/kg over 30 minute IV infusion weekly for 52 weeks, OR initial dose of 8 mg/kg over 90 minutes IV infusion, then 6 mg/kg over 30-90 minutes IV infusion every three weeks for 52 weeks.
  Arms: Her2 positive patients
Drug: T + trastuzumab followed by CEF + trastuzumab — Trastuzumab 4 mg/kg IV for one dose beginning just prior to first dose of paclitaxel.
  Followed by trastuzumab 2 mk/kg IV weekly for 23 weeks Paclitaxel 80 mg/m2 by 1 h IV infusion weekly for 12 wks Followed by 5-Fluorouracil 500 mg/m2 IV on days 1 and 4 Epirubicin 75 mg/m2 IV on day 1 Cyclophosphamide 500 mg/m2 IV on day 1 cycled every 21 days for 4 cycles Trastuzumab 6mg/kg IV every 21 days for 9 cycles to complete 1yr
  Arms: Her2 positive patients
Drug: Dose dense AC followed by T + trastuzumab — Doxorubicin 60 mg/m2 IV day 1 Cyclophosphamide 600 mg/m2 IV day 1 (cycled every 14 days for 4 cycles) Followed by paclitaxel 80 mg/m2 by 1 h IV infusion weekly for 12 wks All cycles are with filgrastim support with trastuzumab 2 mg/kg (4 mg/kg loading dose).
  Following chemotherapy , trastuzumab to continue every 3 weeks at 6 mg/kg for the duration of 1 week.
  Arms: Her2 positive patients
Drug: Dose dense AC followed by T + trastuzumab + pertuzumab — Doxorubicin 60 mg/m2 IV day 1 Cyclophosphamide 600 mg/m2 IV day 1 Cycled every 14 days for 4 cycles Followed by docetaxel 75-100 mg/m2 by 1 h IV infusion weekly for 12 wks All cycles are with filgrastim support with trastuzumab 6 mg/kg (8 mg/kg loading dose with C1) Pertuzumab 420 mg (840 mg loading dose with C1). Following chemotherapy, trastuzumab to continue every 3 weeks at 6 mg/kg for the duration of 1 week.
  Arms: Her2 positive patients
Drug: PTH followed by dose dense AC of FEC — Docetaxel 75-100 mg/m2 by 1 h IV infusion Cycled every 21 days for 4 cycles With Trastuzumab 6 mg/kg IV (8 mg/kg IV loading dose) q3W And Pertuzumab 420 mg IV (840 mg IV loading dose) q 3w +/- pegfilgrastim 6 mg sq on day 2-3,
  Followed by 4 cycles of AC or FEC:
  AC Doxorubicin 60 mg/m2 IV day 1 Cyclophosphamide 600 mg/m2 IV day 1 Cycled every 14 days for 4 cycles with pegfilgrastim 6 mg sq on day 2 FEC 5-Fluorouracil 500 mg/m2 IV on days 1 and 4 Epirubicin 75 mg/m2 IV on day 1 Cyclophosphamide 500 mg/m2 IV on day 1 cycled every 21 days for 4 cycles
  In all of the above mentioned regimens docetaxel might be substituted with paclitaxel as paclitaxel is better tolerated but is expected to have the same efficacy as docetaxel.
  Arms: Her2 positive patients

SUMMARY:
Genomics assays that measure specific gene expression patterns in a patient's primary tumor have become important prognostic tools for breast cancer patients. This study is designed to test the ability of MammaPrint® in combination with TargetPrint®, BluePrint®, and TheraPrint®, as well as traditional pathologic and clinical prognostic factors, to predict responsiveness to neo-adjuvant chemotherapy in patients with locally advanced breast cancer (LABC).

DETAILED DESCRIPTION:
Patients with suspected primary breast cancer on mammography and clinical examination will be assessed for eligibility by having a needle core biopsy to confirm invasive carcinoma.

A fresh unfixed tumor specimen, incisional or core biopsy will be sent to Agendia to determine the MammaPrint risk profile, the BluePrint molecular subtyping profile, the TargetPrint ER, PR and HER2 single gene readout, the 56-geneTheraPrint Research Gene Panel and the additional genes as measured on the whole genome (44k) array.

Surgical Protocol:

1. Determination of nodal status:

   * For clinically node-negative patients: Axillary ultra sound, followed by Sentinel Lymph Node (SLN) biopsy
   * For clinically node-positive patients: ultra sound-guided Fine Needle Aspirate (FNA), followed by core biopsy
2. Neo-adjuvant chemotherapy
3. Definitive surgery:

   * For node-positive patients: lumpectomy, repeat SLN biopsy, Axillary Lymph Node Dissection (ALND)
   * For node-negative patients: lumpectomy, repeat SLN biopsy (optional), no ALND

Response will be measured by pathological Complete Response (pCR) and by centrally assessed Residual Cancer Burden (RCB).

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven invasive breast cancer and no distant metastases and;
* Lymphnode negative and a clinical tumor classification of T2 (≥3.5cm)-T4 or with 1-3 positive lymph nodes and a clinical tumor classification of T2-T4 DCIS or LCIS are allowed in addition to invasive cancer at T2 or T3 level.
* Age ≥ 18 years.
* At least one lesion that can be accurately measured in two dimensions utilizing mammogram, ultrasound, or MRI images to define specific size and validate complete pathologic response.
* Adequate bone marrow reserves (neutrophil count >1.5 x109 /l and platelet count >100 x109/l), adequate renal function (serum creatinine ≤ 1.5 x upper limit of normal) and hepatic function (ALAT, ASAT ≤ 2.5 x upper limit of normal, alkaline phosphatase ≤ 2.5 x upper limit of normal and total bilirubin ≤ 2.0 x upper limit of normal).
* Signed informed consent of the patient

Exclusion Criteria:

* Any patient with confirmed metastatic disease. Patients with inflammatory breast cancer.
* Tumor sample shipped to Agendia with ≤ 30% tumor cells or that fails Quality Assurance or Quality Control criteria.
* Patients who have had any prior chemotherapy, radiotherapy, or endocrine therapy for the treatment of breast cancer.
* Any serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-10; Primary Completion 2016-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Determine the predictive power of chemosensitivity of MammaPrint as measured by pCR. | 6-12 months
Determine the predictive power of chemosensitivity of the combination of MammaPrint and BluePrint as measured by pCR. | 6-12 months

SECONDARY OUTCOMES:
Compare TargetPrint single gene read out of ER, PR and HER2 with local and centralized IHC and/or CISH/FISH assessment of ER, PR and HER2. | Baseline. First study visit.
Identify possible correlations between the TheraPrint Research Gene Panel outcomes and chemoresponsiveness. | 6-9 months
Identify and/or validate predictive gene expression profiles of clinical response/resistance to chemotherapy. | 6-12 months
Compare the three BluePrint molecular subtype categories with IHC-based subtype classification. | Baseline. First study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Cox, MD, Principal Investigator — University of South Florida
Locations (9):
- United States (9):
  - University of South Alabama, Mitchell Cancer Institute, Mobile, Alabama
  - Morton Plant Mease Health Care, Clearwater, Florida
  - University of Miami, Miami, Florida
  - University of South Florida Breast Cancer Program, Tampa, Florida
  - Helen Ellis Memorial Hospital, Tarpon Springs, Florida
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma, Health Sciences Center, Oklahoma City, Oklahoma
  - Texas Health, Plano Cancer Institute, Plano, Texas